CLINICAL TRIAL: NCT01666197
Title: A Randomized, Double-blind, Multi-center, Placebo-controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Diclofenac Potassium 25 mg Tablet Taken Three Times Daily in Subjects With Acute Joint Pain
Brief Title: Efficacy and Safety of Diclofenac Potassium 25 mg Tablet Taken Three Times Daily in Subjects With Acute Joint Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 853-P-401
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Results first posted 2014-03-27 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-03

CONDITIONS: Ankle Sprain
Keywords: Acute Joint Pain
MeSH Terms: conditions — Ankle Injuries | interventions — Diclofenac; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- diclofenac potassium 25 mg tablet (Experimental)
  Interventions: Drug: diclofenac potassium 25 mg tablet
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: diclofenac potassium 25 mg tablet — diclofenac potassium 25 mg tablet
  Arms: diclofenac potassium 25 mg tablet
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of diclofenac potassium 25 mg tablet compared with placebo taken three times a day in subjects with acute ankle sprains under 'in-use' conditions, in particular with regard to pain relief.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years and over.
* Acute sprain of the lateral ankle, Grade I-II, meeting baseline pain intensity level.
* Injury within past 12 hours.

Exclusion Criteria:

* Pain medication was taken within the 6 hours that precede randomization.
* During the past 3 months: Grade I-III sprain of the same ankle.
* During the past 6 months: Grade II-III sprain, any other significant injury (such as fracture or torn ligament), or surgery (except for skin or nails) of the same ankle or foot.
* Pain or instability in the same ankle attributable to previous ankle sprain or any other trauma.
* Ankle sprain attributable to a known disease affecting the ligaments, such as ligament hyperlaxity due to connective tissue disease (e.g., Marfan's syndrome, Down's syndrome, Ehlers-Danlos syndrome).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (4):
  - Investigator, Brühl
  - Investigator, Cologne
  - Investigator, Essen
  - Investigator, Gilching

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Four centers in Germany recruited patients from 22 Aug 2012 to 27 Jan 2013
Period: Overall Study
Arm/Group | Diclofenac Potassium 25 mg Tablet | Placebo
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diclofenac Potassium 25 mg Tablet | Placebo | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.7 (13.4) | 33.2 (12.2) | 32.0 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 47
  Male | 27 | 26 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 50 | 50 | 100
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Pain on Movement
Description: Change on a Visual analog scale from Baseline. Pain on Movement at 48 hours assessed on a 100 mm visual analog scale with anchors at 0="No pain" and 100= "Extreme pain"
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac Potassium 25 mg Tablet | Placebo
Number analyzed (Participants) | 50 | 50
mm | 31.3 (18.8) | 59.2 (12.8)

ADVERSE EVENTS:
Arm/Group | Diclofenac Potassium 25 mg Tablet | Placebo
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 1/50 | 3/50
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diclofenac Potassium 25 mg Tablet (N=50) | Placebo (N=50)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Preliminary agreement between Novartis Consumer Health and the investigator